CLINICAL TRIAL: NCT05952648
Title: HAP/VAP Diagnosis in Critically Ill Septic Patients Using a Multiplex PCR Assay: A Multicenter Randomized Open-Label Trial. THE LIGHTNING STUDY
Brief Title: HAP/VAP Diagnosis in Critically Ill Septic Patients Using a Multiplex PCR Array
Acronym: LIGHTNING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5768
Record Dates: First submitted 2023-07-05; First posted 2023-07-19 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: HAP - Hospital Acquired Pneumonia; VAP - Ventilator Associated Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: Randomized controlled, multicenter, open-label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Film-array Pneumonia Panel Plus group (Experimental): Patients with suspected HAP or VAP in which lower tract respiratory samples are analyzed with new multiplex PCR assay (Film-array Pneumonia Panel Plus)
  Interventions: Procedure: Lower tract respiratory samples; Diagnostic Test: Multiplex PCR assay (Film-array Pneumonia Panel Plus); Diagnostic Test: Lower respiratory tract standard culture; Diagnostic Test: Blood sample standard culture
- Standard culture group (control group) (Active Comparator): Patients with suspected HAP or VAP in which lower tract respiratory samples are analyzed with standard culture
  Interventions: Procedure: Lower tract respiratory samples; Diagnostic Test: Lower respiratory tract standard culture; Diagnostic Test: Blood sample standard culture

INTERVENTIONS:
Procedure: Lower tract respiratory samples — Within 1 hour from HAP or VAP suspicion, quantitative tracheal aspirate or bronchoalveolar lavage will be performed to confirm the diagnosis. Clinicians will be encouraged to perform BAL whenever possible
Diagnostic Test: Multiplex PCR assay (Film-array Pneumonia Panel Plus) — The lower tract respiratory samples will be analyzed with Multiplex PCR assay (Film-array Pneumonia Plus).
  Arms: Film-array Pneumonia Panel Plus group
Diagnostic Test: Lower respiratory tract standard culture — The lower tract respiratory samples will be analyzed using convention microbiological methods (including conventional Gram stain and semiquantitative culture on both selective/differential and screening agar media)
Diagnostic Test: Blood sample standard culture — When HAP or VAP are suspected, blood samples from peripheral vein will be collected and analyzed with conventional microbiological methods

SUMMARY:
Multicenter, randomized, controlled, open-label trial to assess if semiquantitative multiplex PCR assay, as compared to conventional microbiology, can reduce the percentage of patients without microbiological diagnosis in the first 24 hours from HAP/VAP suspicion, thus allowing early de-escalation.

DETAILED DESCRIPTION:
Hospital-acquired pneumonia and ventilator-associated pneumonia are leading cause of morbidity and mortality in Intensive Care Unit due to the underlining clinical conditions of critically ill patients and the high rate of multidrug resistance among causative agents.

In patients with sepsis and septic shock, early and appropriate antibiotics are essential for improving clinical outcome, often requiring the use of broad-spectrum combinations.

The optimal use of antimicrobials is part of current implementation programs aimed to reduce the administration of not-necessary antibiotics, the bio-ecologic pressure and the possible side effects .

In this context the application of rapid, molecular microbiological tests on respiratory samples is of overwhelming interest, due to the potential of reducing the time to inappropriate antibiotic therapy and of prompting de-escalation.

During last years a new Multiplex PCR Assay for pneumonia diagnosis (Film-Array Pneumonia Panel Plus, BioFire, Salt Lake City, UT, USA) has been implementing in the clinical practice, showing very high rates of negative and positive predictive values.

The hypothesis is that molecular test on lower respiratory tract samples may reduce the time to microbiological diagnosis, thus allowing early antibiotic de-escalation.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of HAP/VAP (clinical/radiological/laboratory criteria);
* Availability to perform tracheal aspirates or broncoalveolar lavage within 1 hour from clinical suspicion
* Life expectancy ≥ 48 hours
* Signed written informed consent.

Exclusion Criteria:

* Pregnancy,
* Concomitant participating in other interventional trial
* Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients without microbiological diagnosis of HAP/VAP within the first 24 hours | 24 hours
  Proportion of patients where a microbiological diagnosis of HAP/VAP is not avaiable within the first 24 hours

SECONDARY OUTCOMES:
Rate of antibiotic de-escalation as a consequence of microbiological results | 4 days
  Proportion of patients in which antibiotic therapy has been modified from broad-spectrum empirical to targeted, due to microbiological results
Time to antibiotic de-escalation and optimal therapy | 4 days
  Period of time from empirical antibiotic therapy initiation to modification due to microbiological results
Mechanical Ventilation free-days | 14 and 28 days
  Number of days from enrollment in which the patients is not mechanically ventilated
Rate of MDR infection | 28 days
  Proportion of patients who suffered from infection caused by multidrug resistant germ
Lenght of intensive care unit stay | 60 days
  Period of time from enrollment in which the patient is admitted to the intensive care unit
Lenght of hospital stay | 60 days
  Period of time from enrollment in which the patient is admitted to the hospital
In-Intensive care unit mortality | 28 days and 60 days
  All-cause mortality, assessed during ICU stay
28 days and 60 days mortality | 28 days and 60 days
  All-cause mortality
SOFA score | 14 days
  Measured SOFA score after 2,3,7 and 14 days from enrollment
Diagnostic concordance | 4 days
  Proportion of patients in the interventional group, in which microbiological diagnosis is concordant when assessed with PCR array and standard culture
Adverse event | 28 days
  Proportion of patients in which any adverse event is registered
In-Hospital mortality | 28 days and 60 days
  All-cause mortality, assessed during Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro De Pascale, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS; Massimo Antonelli, MD, Study Chair — Fondazione Policlinico A. Gemelli IRCCS
Locations (4):
- Italy (4):
  - S. Orsola Research Hospital, Bologna
  - Ospedale Careggi, Florence
  - Modena Policlinico, Modena
  - Fondazione Policlinico Universitario "A. GEMELLI" IRCCS, Roma